CLINICAL TRIAL: NCT05720091
Title: A Study to Evaluate the Substance Balance of [14C] ZX-7101A in Healthy Adult Male Subjects in China
Brief Title: Substance Balance Study of [14C]ZX-7101A in Healthy Adult Male Subjects in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX-7101A-204
Record Dates: First submitted 2023-01-16; First posted 2023-02-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZX-7101A (Experimental)
  Interventions: Drug: ZX-7101A 80mg

INTERVENTIONS:
Drug: ZX-7101A 80mg — a drug to treatment influenza in Chinese adults

SUMMARY:
The objectives of this substance balance study in healthy Chinese adult male subjects are to obtain human radioactivity recovery data and major excretion pathways, and to obtain pharmacokinetics of total radioactivity in plasma, and to identify major metabolites in the radiometabolite spectrum. The main questions it aims to answer are:

* Quantitative analysis of total fecal and urine radioactivity in healthy subjects after oral administration of [14C]ZX-7101A to obtain human radioactive recovery data and main excretion routes.
* Pharmacokinetics of total activity in whole blood and plasma, and distribution of total activity in whole blood and plasma are quantitatively analyzed after oral administration of [14C]ZX-7101A in healthy subjects.
* Quantitative analysis of the radioactive metabolites in plasma, urine and feces of healthy subjects with once [14C]ZX-7101A orally administration, identification of the main metabolites of the radioactive metabolites (close to or greater than 10% of the total radioactive AUC in plasma), and determination of the main biotransformation and elimination pathway of ZX-7101A.

ELIGIBILITY:
Inclusion Criteria:

* The body mass index (BMI) is 19.0 to 26.0 kg/m2 (including the cut-off), and the subject must weigh no less than 50kg.
* Before the test, fully understand the test content, process and possible adverse reactions, and voluntarily sign the informed consent.

Exclusion Criteria:

* People with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product.
* Subjects with a pre-existing or present history of metabolic, liver, kidney, hematological, pulmonary, cardiovascular, gastrointestinal, urinary, endocrine, neurological, or psychiatric disease with clinical manifestations that the investigator deems unsuitable for participation in this study.
* Hemorrhoids or perianal disease with regular/ongoing blood in the stool, irritable bowel syndrome, inflammatory bowel disease.
* Screening for novel coronavirus infection: Those who are positive for novel coronavirus nucleic acid.
* Physical examination, vital signs, routine laboratory examination , thyroid function, chest CT, abdominal B-ultrasound and other tests were abnormal with clinical significance.
* Estimated glomerular filtration rate <90 mL/min/1.73 m2 (see Appendix 1 for eGFR formula).
* Resting corrected QT interval (QTcF) ≥450ms, QRS≥120ms obtained by 12-lead electrocardiogram (ECG).
* Any conditions that may affect drug absorption, such as gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy, history of inflammatory bowel.
* Previous history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmias, torsional ventricular tachycardia, ventricular tachycardia, atrioventricular block, history of prolonged QT syndrome, or symptoms of prolonged QT syndrome, and family history (indicated by genetic evidence or by sudden cardiac death at a young age in a close relative).
* Major surgery or surgical incision not fully healed within 6 months prior to the screening period; Major surgery includes, but is not limited to, any surgery where there is a significant risk of bleeding, prolonged period of general anesthesia, or open biopsy or significant traumatic injury.
* Use of any P-gp inducer or inhibitor within 30 days prior to the screening period; Have used any prescription drugs or Chinese herbs within 14 days prior to the screening period.
* Those who consumed more than 14 units of alcohol per week (1 unit of alcohol =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine) within the six months prior to screening or tested positive for alcohol breath at the screening.
* Smokers who smoked more than 5 cigarettes a day or habitually used nicotine-containing products within the 3 months before screening and could not quit during the trial period.
* Subjects who tested serologically positive for antibodies to syphilis (Treponema pallidum), hepatitis B surface antigen or E antigen, hepatitis C virus antibody or human immunodeficiency virus antibody during the screening period.
* Those who had lost blood or donated 400 mL in the 3 months prior to the screening period or donated >200 mL within 4 weeks or planned to donate blood during the study period.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery of total radioactive material in urine and feces | From 1 days before medication to 22 days after medication
  The total radioactivity in excreta of healthy subjects after oral administration of [14C]ZX-7101A
Cmax of total radioactivity in plasma | From 1 days before medication to 22 days after medication
  The peak concentration of ZX-7101A after oral administration of [14C]ZX-7101A in healthy subjects
AUC of total radioactivity in plasma | From 1 days before medication to 22 days after medication
  The area under curve of ZX-7101A after oral administration of [14C]ZX-7101A in healthy subjects

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From medication to 22 days after medication
  The Treatment-Related Adverse Events of ZX-7101A will be evaluated by the change of vital signs, electrocardiogram (P Wave, QRS Complex, QT Interval), physical examination, and Laboratory test compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: liyan Miao, doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No